CLINICAL TRIAL: NCT06636500
Title: A Phase 1, Single and Multiple Ascending Dose and Food Effect Study of CG001419 Administered Orally to Evaluate Safety, Tolerability and Pharmacokinetics in Healthy Subjects
Brief Title: A Phase 1 Study of CG001419 Administered Orally in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cullgen Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CG001419-101
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteer Study; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CG001419 (Experimental): Part A: Single ascending dose cohorts; food effect cohort; Part B: Multiple ascending dose cohorts
  Interventions: Drug: CG001419
- Placebo (Placebo Comparator): Part A: Single ascending dose cohorts; Part B: Multiple ascending dose cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CG001419 — Oral doses
  Arms: CG001419
Drug: Placebo — Oral doses
  Arms: Placebo

SUMMARY:
This is a dose finding study of CG001419, administered as a single dose, with or without food, and as multiple doses. CG001419 is being tested in healthy volunteers in this trial with the goal of eventually developing the drug for patients with pain if it is found to be safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Cis-male and cis-female subjects must be 18-65 years, inclusive, at the time of signing the informed consent form (ICF).
* Subjects who are in good general health according to the judgment of the investigator per local guidance, eg, with no clinically relevant abnormalities based on medical history, physical examinations, neurological examinations, clinical laboratory evaluations (hematology and clinical chemistry), vital signs, and 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, would affect subject safety.
* Subjects who have a body mass index (BMI) of 18-32 kg/m2 (inclusive) at screening.
* Male subjects are eligible to participate if they are permanently sterile by vasectomy (at least 6 months), or agree to the following during the study and for at least 90 days after the last dose of study drug:

  1. Refrain from donating sperm

     AND, either:
  2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent OR
  3. Agree to use a male condom (contraception/barrier) and should also be advised of the benefit for a female partner to use an acceptable, highly effective method of contraception (of low user dependency or is user dependent), as a condom may break or leak when having sexual intercourse 5. Female subjects are eligible to participate if they are not pregnant or breastfeeding and fall under 1 of the following criteria:

  <!-- -->

  1. Women of childbearing potential (WOCBP), defined as women physiologically capable of becoming pregnant, must have a negative serum pregnancy test at the Screening visit and a negative urine pregnancy test on Day -1; WOCBP must agree to be abstinent from heterosexual intercourse or use an acceptable, highly effective contraceptive method (of low user dependency or is user dependent) from Screening and not donate eggs until 30 days after the last dose of the study drug.

     OR
  2. Menopausal women must have an elevated serum follicle-stimulating hormone level (FSH >40 IU/mL) level at Screening; if the FSH is not elevated, they are considered to be of childbearing potential (unless permanently sterile).

Exclusion Criteria:

* Clinically significant infection and/or cardiovascular, hematological, renal, hepatic, pulmonary (except recovered childhood asthma), endocrine, reproductive, gastrointestinal, immunological, dermatological, neurological (except migraine), or psychiatric (except depression, which was potentially medicated in the past but didn't require hospitalization) diseases, which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the investigator, unacceptably increase the subject's risk if he/she were to participate in the study.
* History of neuropathy and/or any neurosensory symptoms in the feet or hands.
* Unable to ingest a high-fat meal, such as those who are lactose intolerant (only for subjects in the FE part and if recommended, MAD part too)
* History of disorders that affect gastrointestinal transit time (eg, short bowel syndrome, gastroparesis, irritable bowel syndrome, inflammatory bowel diseases, history of gastric bypass
* Use of prescription drugs, over-the-counter drugs (other than acetaminophen and ibuprofen), herbal medications, or vitamin supplements within 7 days or 5 half-lives, whichever is longer, prior to dosing and antibiotics and systemic steroids within 30 days prior to dosing. Oral contraceptives are permitted. The sponsor, after consulting medical monitor may allow exceptions only if the medication's administration is deemed unlikely to impact the PK results.
* Past or current history or evidence of drug or alcohol abuse, alcohol consumption exceeding 5 units of alcohol on an average per day (1 unit of alcohol = 150 mL of wine, 360 mL of beer, or 45 mL of alcohol 40%). Use of any non-marijuana illicit drugs (e.g., cocaine, phencyclidine) within 6 months of Screening.
* Donation of over 500 mL of blood within 8 weeks prior to Screening.
* In the opinion of the investigator the subject is unlikely to comply with the study procedures, restrictions, and requirements and is not suitable for entry into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple ascending oral doses of CG001419 in healthy subjects | Up to 7 days of dosing
  Safety and tolerability based on adverse events (AEs)

SECONDARY OUTCOMES:
To further characterize the PK of CG001419 in healthy subjects | Up to 7 days of dosing
  Cmax
To further characterize the PK of CG001419 in healthy subjects | Up to 7 days of dosing
  Tmax
To further characterize the PK of CG001419 in healthy subjects | Up to 7 days of dosing
  Area under the concentration curve from 0 to last (AUC0-last)
To further characterize the PK of CG001419 in healthy subjects | Up to 7 days of dosing
  Area under the concentration curve from 0 to infinity (AUC0-inf)
To further characterize the PK of CG001419 in healthy subjects | Up to 7 days of dosing
  Elimination rate constant (λz)
To further characterize the PK of CG001419 in healthy subjects | Up to 7 days of dosing
  Terminal elimination half-life (t1⁄2)
To further characterize the PK of CG001419 in healthy subjects | Up to 7 days of dosing
  Apparent oral clearance (CL/F)
To further characterize the PK of CG001419 in healthy subjects | Up to 7 days of dosing
  Apparent volume of distribution (Vd/F)

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
This is a healthy volunteer study being conducted to define the safety profile of the drug. This study is not exploring the activity of our drug in the target indication population (patients with pain). As such, we do not believe there is utility for sharing deidentified IPD from this trial with other researchers.